CLINICAL TRIAL: NCT05235516
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate AK104 Combined With Chemoradiotherapy For The Treatment of Locally Advanced Cervical Cancer
Brief Title: A Study of AK104/Placebo Combined With Chemoradiotherapy For The Treatment of Locally Advanced Cervical Cancer
Acronym: AK104-305
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK104- 305
Record Dates: First submitted 2022-01-20; First posted 2022-02-11 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Cervical Carcinoma
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment arm (Experimental)
  Interventions: Drug: AK104; Radiation: EBRT; Radiation: BT; Drug: cisplatin
- placebo arm (Placebo Comparator)
  Interventions: Radiation: EBRT; Radiation: BT; Drug: cisplatin; Drug: Placebo

INTERVENTIONS:
Drug: AK104 — q3w iv
  Arms: treatment arm
Radiation: EBRT — 45-50.4Gy
Radiation: BT — ≥80Gy
Drug: cisplatin — qw iv
Drug: Placebo — q3w iv
  Arms: placebo arm

SUMMARY:
This study is to evaluate the efficacy and safety of AK104 plus concurrent chemoradiotherapy compared to placebo plus concurrent chemoradiotherapy in participants with locally advanced cervical cancer

ELIGIBILITY:
Inclusion Criteria:

1. signs the written informed consent form
2. ECOG 0-1
3. Life expectancy ≥ 3 months.
4. The histological types include squamous cell carcinoma,adenocarcinoma, or adenosquamous cell carcinoma;
5. Locally advanced cervical cancer (LACC): The International Federation of Gynecology and Obstetrics (FIGO) 2018 Stage 3A-4A
6. At least one measurable tumor lesion per RECIST v1.1
7. Adequate organ function as assessed in the laboratory tests

Exclusion Criteria:

1. Subjects with other histopathological types of cervical cancer, such as small cell carcinoma, sarcoma, etc.
2. FIGO 2018 IVB
3. Subjects who had previously undergone total hysterectomy
4. Subjects who cannot receive brachytherapy
5. Subjects with other active malignancies within 2 years prior to randomization
6. Clinically significant hydronephrosis that cannot be relieved by nephrostomy or ureteral stenting as judged by the Investigator
7. Any prior treatments targeting the mechanism of tumor immunity, such as immune checkpoint inhibitors (e.g., anti-PD-1 antibody, anti-PDL1 antibody, anti-CTLA-4 antibody, etc.), or therapy against immune costimulatory factors (e.g., antibodies directed against ICOS, CD40,CD137, GITR, OX40 targets, etc).
8. Subjects who require systemic treatment with glucocorticoid (>10 mg/day of prednisone or equivalent glucocorticoid) or other immunosuppressive agents within 14 days prior to randomization;
9. Major surgical treatment, open biopsy or significant trauma within 4 weeks prior to randomization; or elective major surgical treatment required during the study
10. Use of live vaccines within 4 weeks prior to randomization
11. Active or potentially recurrent autoimmune disease
12. Known primary or secondary immunodeficiencies, including testing positive for human immunodeficiency virus (HIV) antibodies
13. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
14. Known history of interstitial lung disease or non-infectious pneumonitis
15. Pregnant or lactating women.
16. Any condition that, in the opinion of the Investigator, may result in a risk when receiving the study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) by investigator(INV) | 54 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1 and/or biopsy

SECONDARY OUTCOMES:
PFS rate at month 36 | 36 months
  PFS rate at month 36
Overall Survival(OS) | 5 years
  OS is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Ph.D, Principal Investigator — Sun Yat-sen University; Yang Xiang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan cancer hospital, Changsha, Hunan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Second University Hospital, Chengdu, Sichuan
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided